CLINICAL TRIAL: NCT00563329
Title: Smoking Reduction Intervention for Smokers Not Willing to Quit Smoking: a Randomised Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: UW 03-103 T/103; HARECCTR0500051
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Smoking Cessation
Keywords: Smokers who are not willing to quit in the near future but intend to reduce smoking
MeSH Terms: conditions — Smoking Cessation

INTERVENTIONS:
Procedure: Reduction Intervention + Adherence Intervention
Behavioral: Reduction Intervention
Procedure: control

SUMMARY:
The aims of this study are (1) to examine the effect of smoking reduction intervention (reduction counseling and nicotine replacement therapy, NRT) (a) on smoking cessation and (b) on reducing daily cigarette consumption among smokers not willing to quit smoking but want to reduce smoking, and (2) to examine the effect of adherence intervention in producing a higher (a) adherence rate, (b) reduction rate, and (c) quit rate.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Ethnic Chinese male or female
* Smokes at least 2 cigarettes per day
* Have no intention to quit in the near future
* Intends to reduce smoking in the next 7 days
* Has no contraindication to NRT

Exclusion Criteria:

* Subjects who are psychologically or physically unable to communicate
* Children and teenagers (age below 18)
* Pregnant or intention to become pregnant within the next 6 months
* Those on regular psychotropic medications and in the presence of any serious health problems that may make them unsuitable for using NRT, such as recent stroke, palpitation, or other life threatening conditions

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 3826 (Estimated)
Dates: Start 2004-10; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
quit rate | 6 months
Reduction Rate (reduction of cigarette consumption by at least 50% compared with baseline) | 6 months
Adherence Rate to NRT | 4 weeks

SECONDARY OUTCOMES:
Validated quit rate (by measuring exhaled CO and urinary cotinine level) | 6 months
Quit rate without validation | 1 month
self-reported use of NRT for at least 4 weeks or 8 weeks, without cotinine validation | 1 month / 3 month

CONTACTS AND LOCATIONS:
Overall Officials: TH Lam, Prof, Principal Investigator — Department of Community Medicine, Faculty of Medicine, The University of Hong Kong
Locations (3):
- China (3):
  - HAHO, Hong Kong
  - Hong Kong Council on Smoking and Health, Hong Kong
  - The University of Hong Kong, Hong Kong